CLINICAL TRIAL: NCT03774095
Title: Effects of Pine Nut and Olive Oil as FFA1/FFA4 and GPR119 Agonists on Glucose Tolerance in Healthy Overweight or Obese Subjects
Brief Title: Effect of Dietary Oils as G-protein-coupled Receptor Agonists on Glucose Tolerance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karina Vejrum Sørensen (Other)
Responsible Party: Sponsor-Investigator, Karina Vejrum Sørensen, MSc, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PINO 5
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: incretins; Fat metabolites; Free fatty acid receptors; G-protein-coupled receptors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: Cross-over study of 3 interventions; 1) no oil intake, 2)6g hydrolyzed pine nut oil and 3) combined intake of 3g hydrolyzed pine nut oil and 3g olive oil 30 minutes prior to an 6-hours oral glucose tolerance test (75g glucose).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No oil (No Intervention): 6-hour oral glucose tolerance test
- Hydrolyzed pine nut oil (Active Comparator): 6g hydrolyzed pine nut oil in delayed release capsules given 30 min prior to an 6-hour oral glucose tolerance test
  Interventions: Dietary Supplement: Hydrolyzed pine nut oil
- Hydrolyzed pine nut oil and olive oil (Active Comparator): 3g hydrolyzed pine nut oil and 3g olive oil in delayed release capsules given 30 min prior to an 6-hour oral glucose tolerance test
  Interventions: Dietary Supplement: Hydrolyzed pine nut oil and olive oil

INTERVENTIONS:
Dietary Supplement: Hydrolyzed pine nut oil — Given 30 min prior to oral glucose tolerance test
  Arms: Hydrolyzed pine nut oil
Dietary Supplement: Hydrolyzed pine nut oil and olive oil — Given 30 min prior to oral glucose tolerance test
  Arms: Hydrolyzed pine nut oil and olive oil

SUMMARY:
Agonistic activation of fat metabolite responsive G-protein-coupled receptors (GPCR) has been linked to improved glucose metabolism through increased glucose-stimulated-insulin-secreting (GSIS) and incretin release, improved insulin sensitivity and reduced low grade inflammation. In vitro studies have demonstrated that pinolenic acid (20% of pine nut oil) is a potent dual agonist of two GPCRs: free fatty acid receptor-1 (FFA1, formerly GPR40) and free fatty acid receptor-4 (FFA4, formerly GPR120). Moreover, pinolenic acid was able to improve glucose tolerance in mice. G-protein-coupled receptor-119 (GPR119) is known to be activated by the monoacylglycerol: 2-oleoylglycerol (2OG), which is a glycerol molecule attached to oleic acid in the second position. Olive oil contains 61-80% oleic acid, and under digestion 2OG is produced. 2OG has been shown to stimulate GLP-1 release in humans and interestingly, it has recently been suggest that simultaneous activation of GPR119 and FFA1 acts in synergy and enhances enteroendocrine GLP-1 secretion more than the summarized individual agonistic activation. However, this remains to be evaluated in humans. The investigators hypothesize that a combination of pinolenic acid and 2OG administered in delayed release capsules will act in synergy and enhance 1) GLP-1 secretion by stimulating FFA1/FFA4 and GPR119 on enteroendocrine cells causing improved GSIS and increased satiety and 2) enhance GSIS by directly stimulating FFA1 and GPR119 on beta-cells.

Study aim: To investigate the acute effects of pinolenic acid combined with 2OG (olive oil) versus pinolenic acid alone on changes in glucose tolerance, insulin, GLP-1, GIP and ghrelin secretion, appetite and gastrointestinal tolerability in overweight and obese healthy humans.

DETAILED DESCRIPTION:
During the last decade, several G protein-coupled receptors (GPCR) that respond to dietary lipid metabolites including free fatty acids (FFAs) have been discovered. These receptors have been implicated in metabolic processes and inflammation. Consequently, several of the receptors have attracted interest as potential targets for the treatment of metabolic and inflammatory diseases, including obesity and type 2 diabetes (T2D).

Free fatty acid receptor 1 (FFA1 or GPR40) is activated by long-chain FFAs and is highly expressed in pancreatic β-cells, where it increases glucose-stimulated insulin secretion (GSIS). FFA1 is also expressed on intestinal enteroendocrine cells, where it promotes secretion of incretin hormones such as glucagon like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP). GLP-1 is highly interesting for treatment of obesity and T2D because of its ability to increase GSIS, enhance β-cell growth, increase insulin sensitivity, reduce gastric motility, increase satiety and reduce body weight. The published phase II clinical trial with the selective FFA1 agonist TAK-875 demonstrated high efficacy in reducing plasma glucose without increased incidence of hypoglycemia, and has caused considerable interest in the receptor as a new target for treatment of type 2 diabetes. Free fatty acid receptor 4 (FFA4 or GPR120) is activated by unsaturated long-chain FFAs and is expressed in the gastrointestinal system and adipose tissue. It is reported to promote GLP-1 secretion from intestinal cells, to counteract inflammation and to increase insulin sensitivity in adipose tissue. Notably, dysfunctional FFA4 was recently connected to the development of obesity in both mice and humans. This has considerably increased the interest on the receptor as a target for obesity and metabolic diseases.

Another GPCR receptor: G-protein-coupled receptor-119 (GPR119), which reacts to different degradation products of triacylglycerol including monoacylglycerols, has similar functions as FFA1 and FFA4. It is also expressed in enteroendocrine cells in the gastrointestinal tract and on pancreatic β-cells, where it stimulates GLP-1 secretion and GSIS, respectively.

In summary, these receptors are expressed in different tissues in the body where they potentially can affect metabolic and inflammatory conditions such as type 2 diabetes and obesity.

Prior to this study, an in in vitro screening of 36 relevant FFAs and their ability to act as FFA1 and FFA4 agonists was carried out to identify the most potent naturally occurring dual FFA1/FFA4 agonist for clinical studies. Of these, the polyunsaturated fatty acid, pinolenic acid showed the highest efficacy and a good potency on both receptors, and was therefore selected for further studies.

To further support this choice, the effect of pinolenic acid was tested using a small dose (100 mg/kg) given 30 min prior to an oral glucose tolerance test (OGTT) in mice. Convincingly, purified pinolenic acid significantly improved glucose tolerance by reducing OGTT glucose levels when compared to control (corn oil). The efficacy was similar to that obtained with a pharmaceutical selective FFA1 agonist (TUG-905). Pinolenic acid is a fatty acid contained in Siberian Pine nuts, Korean Pine nuts and the seeds of other pines. The highest percentage of pinolenic acid (~20%) is found in Siberian Pine nuts and the oil produced from them. Korean Pine nut oil given as hydrolyzed FFAs, but not as triglycerides, has been reported to increase secretion of GLP-1 and decrease appetite in overweight females. This supports the indication that purified pinolenic acid may be superior in improving glucose metabolism.

GPR119 is activated by different endogen ligands, one of them being the monoacylglycerol 2-oleoylglycerol (2OG), which is a glycerol molecule attached to oleic acid in the second position. Olive oil contains 61-80% oleic acid, and under digestion of 5 ml olive oil, approximately 2g 2OG is produced. 2OG has been shown to stimulate GLP-1 release in humans and interestingly, it has recently been suggest that simultaneous activation of GPR119 and FFA1 acts in synergy and enhances enteroendocrine GLP-1 secretion more than the summarized individual agonistic activation. However, this remains to be evaluated in humans.

Roux-en-Y gastric bypass (RYGB) surgery, used to treat severe obesity, frequently results in immediate beneficial effects on glucose metabolism in type 2 diabetes, often with complete remission. These effects are in part independent of weight loss, but may be explained by a significant increase in GLP-1 levels immediately after surgery. Thus, it appears that the effect depends on the delivery of nutrients to the lower parts of the intestine. Fat metabolites are normally rapidly absorbed in the upper parts of the gastrointestinal tract. It is therefore possible that the RYGB effects are partly due to enteroendocrine stimulation of FFA1, GPR119 and perhaps FFA4 by direct nutrient delivery, that is, delivery of fat metabolites to the lower intestines. A hypothesis to be investigated in this study is that the delivery of pinolenic acid and 2OG to the lower intestines can mimic the beneficial effects observed after RYGB with less expense and fewer adverse effects.

Delivery of nutrients beyond the proximal small intestine can be achieved by the use of delayed release capsules. The potential positive effect of this principle was recently reported in a small cohort of patients with T2D. Where, delivery of small amounts of lauric acid (a C12 fatty acid) to the distal gut using enteric-coated pellets stimulated GLP-1 secretion and lowered postprandial glucose levels in response to meals. No chronic effects where tested in this study. Although not suggested by the authors, the increased release of GLP-1 could involve direct stimulation of FFA1 and/or FFA4 by lauric acid in the distal gut.

Hypotheses: As described, the expression of FFA1, FFA4 and GPR119 on intestinal enteroendocrine cells and pancreatic beta-cells has been linked to 1) increased secretion of GLP-1 and GIP hence the incretin-mediated increase in GSIS and 2) a direct positive effect on GSIS. The investigators hypothesize that a combination of pinolenic acid and 2OG administered in delayed release capsules will act in synergy and 1) enhance GLP-1 secretion by stimulating FFA1/FFA4 and GPR119 on enteroendocrine cells causing improved GSIS, 2) enhance GSIS by directly stimulating FFA1 and GPR119 on beta-cells and 3) increase satiety.

To test the hypotheses, the aim of this project is to investigate the acute effect of pinolenic acid (hydrolyzed pine nut oil) combined with 2OG (olive oil) versus pinolenic acid (hydrolyzed pine nut oil) alone on glucose tolerance, insulin, GLP-1, GIP and ghrelin secretion, appetite and gastrointestinal tolerability in overweight and obese healthy humans.

ELIGIBILITY:
Inclusion Criteria: body mass index (BMI) of 27.5-40 kg/m2, normal glucose tolerance (two hours OGTT plasma glucose ≤ 7.8 mmol/l), normal blood pressure and normal screening blood samples (kidney and liver function, lipids and hematology) and written informed consent -

Exclusion Criteria:any chronic disease including past gastrointestinal diseases or gastrointestinal surgery, first degree relatives with diabetes, food allergies of relevance, need for prescriptive medicine, smoking, body weight changes (> 3 kg within three month prior), intake of dietary supplements (<1 month prior) or any type of restrictive diet for example calorie restriction, vegan diet etc.

-

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Glucose | 6 hours
  Glucose area under the curve
Insulin | 6 hours
  Insulin area under the curve
C-peptide | 6 hours
  C-peptide area under the curve
GLP-1 | 6 hours
  GLP-1 area under the curve
GIP | 6 hours
  GIP area under the curve
Ghrelin | 6 hours
  Ghrelin area under the curve
Appetite | 6 hours
  Appetite is measured by the use of Visual analog scales. Respondents specify their level of agreement to a statement on hunger, satiety, fullness, prospective food consumption and thirst by indicating a position along a continuous 100 mm line between two end-points (0 and 100 mm) which represent the extreme feelings related to the statement. In example: How hungry do you feel? 0mm represents: Not hungry at all and 100 mm represents: I have never been hungrier.
Gastrointestinal tolerability | 24 hours
  Gastrointestinal tolerability is measured by the use of Visual analog scales. Respondents specify their level of nausea, flatulence, abdominal pain, diarrhea and constipation by indicating a position along a continuous 100 mm line between two end-points (0 and 100 mm) which represent the extreme feelings related to the symptom in question. In example: Have you been constipated? 0mm represents: No,not at all and 100 mm represents: Yes, severely.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Hø, MD, Principal Investigator — Odense University Hospital/ University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark